CLINICAL TRIAL: NCT05402514
Title: Digitally Delivered Exercise and Education Treatment for Shoulder Pain: 3 Months Follow-up
Status: Completed | Type: Observational
Sponsor: Joint Academy (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: Shoulder3months
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Shoulder Pain; Subacromial Pain Syndrome
Keywords: Shoulder pain; Rehabilitation; Physical Therapy Modalities; Telerehabilitation; Exercise therapy; Patient education as Topic
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Digitally delivered exercise and education treatment Joint Academy — The Joint Academy® (www.jointacademy.com) program for people with subacromial shoulder pain consist of two daily distributed and progressively adaptable exercises there are delivered through the app as videos with subtitles. Patient education is provided 2-3 times per week as short lessons in the app with a quiz following the text to ensure that the information is properly understood by the patients. An individual physical therapist is assigned to each patient with compulsory telephone or video consultations at the start of the treatment, at 6 weeks and at 3 months. An asynchronous chat function with the physical therapist is available during the treatment period as well as a peer support chat.

SUMMARY:
The overall aim of this project is to describe changes in pain and perceived shoulder dysfunction in patients with subacromial shoulder pain, following 3 months of digitally delivered first-line treatment containing exercise and patient education with support of a licensed physical therapist.

The intervention, a digital first-line treatment for subacromial shoulder pain is a part of the public healthcare system in Sweden and all residents in the country can access the treatment. The treatment program is based on the existing evidence for treating subacromial shoulder pain and is inspired by specific exercises that have been documented to reduce the need for surgery in the patient group. The program focuses on strengthening the rotator cuff and the muscles stabilizing the scapula. The intervention procedure is similar to previous digital treatments by the same digital care provider and is thoroughly described in previous studies.

DETAILED DESCRIPTION:
Musculoskeletal conditions are identified by the Global Burden of Disease Study as a leading cause of global morbidity. Estimates of the need for rehabilitation services show that at least one in every three people in the world needs rehabilitation at some point in their life course. As disability becomes an increasingly large component of disease burden and health expenditure, greater research and development investment is needed to identify new, more effective intervention strategies.

Traditional face-to-face interventions present barriers, such as limited access and lack of flexibility, which may limit the patients' adherence with the interventions. Digital delivery of the management program may be one way of overcoming such barriers. Telerehabilitation has been successfully implemented and compared to conventional treatments, where adherence to digital treatment has been shown to be associated with an improvement in function and pain in a variety of musculoskeletal(MSK) conditions. The evidence for digital delivered rehabilitation for shoulder pain indicates that it may be a promising way of delivering treatment for the patient group but is still at an early stage and more research is needed.

The overall aim of this project is to describe changes in pain and perceived shoulder dysfunction in patients with subacromial shoulder pain, following 3 months of digitally delivered first-line treatment containing exercise and patient education. A further aim is to compare changes in outcomes between patients with different demographics, and health- and treatment related factors.

The study will be an observational, registry-based longitudinal study with consecutively recruited participants. Socio-demographic data will be collected at baseline including variables such as age, sex, weight, height, highest level of education reached and current job status. All data will be collected through digitally delivered questionnaires in the app at baseline and 3 months besides pain levels, which will be reported weekly until treatment week 6. All outcomes will be self-assessed through the digital program interface. The study will be presented in accordance to the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Subacute or long term subacromial pain

Exclusion Criteria:

* acute pain caused by trauma within the past 3 months that has not yet been physically examined
* signs of acute infection
* suspected undiagnosed malignancy
* radiculopathy from the neck
* shortness of breath or chest pain combined with shoulder pain

Patients excluded from the program will be welcomed back into the treatment after a physical visit if medical professional conclude that they are eligible for physical therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients eligible for the digital first-line treatment program for subacromial shoulder pain with given informed consent will be included in the study. General marketing through different media channels, the company website and word of mouth will be used to recruit patients for the treatment. Patients will not be required to have a doctor or physical therapist referral to enter the treatment. Patients without a prior diagnosis will be assessed and diagnosed by a physical therapist per phone or video call.
Sampling Method: Non-Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Pain Numeric Rating Scale (NRS) | Weekly changes and baseline to 3 month follow-up
  Shoulder pain will be assessed using NRS with the instructions "Mark on the scale your average pain from your shoulder in the past week", followed by a 0-10 scale where 0 is described as "No pain" and 10 described as "Unbearable". Higher scores means worse outcome.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Baseline and follow-up after 3 months
  The self administered Shoulder Pain and Disability Index (SPADI) will be collected at baseline and at 3 months to assess shoulder function. The questionnaire contains 13 items and the score is expressed as percentage where 0 is the best score and 100 the worst score. A higher score means more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Leif E Dahlberg, Professor, Study Director — Arthro Therapeutics /Joint Academy
Locations (1):
- Joint Academy, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmgren T, Hallgren HB, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. Br J Sports Med. 2014 Oct;48(19):1456-7. doi: 10.1136/bjsports-2014-e787rep. PMID 25213604
- [Background] Lee AC. COVID-19 and the Advancement of Digital Physical Therapist Practice and Telehealth. Phys Ther. 2020 Jul 19;100(7):1054-1057. doi: 10.1093/ptj/pzaa079. No abstract available. PMID 32343836
- [Background] Gohir SA, Eek F, Kelly A, Abhishek A, Valdes AM. Effectiveness of Internet-Based Exercises Aimed at Treating Knee Osteoarthritis: The iBEAT-OA Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e210012. doi: 10.1001/jamanetworkopen.2021.0012. PMID 33620447
- [Background] Pieters L, Lewis J, Kuppens K, Jochems J, Bruijstens T, Joossens L, Struyf F. An Update of Systematic Reviews Examining the Effectiveness of Conservative Physical Therapy Interventions for Subacromial Shoulder Pain. J Orthop Sports Phys Ther. 2020 Mar;50(3):131-141. doi: 10.2519/jospt.2020.8498. Epub 2019 Nov 15. PMID 31726927
- [Background] Haik MN, Alburquerque-Sendin F, Moreira RF, Pires ED, Camargo PR. Effectiveness of physical therapy treatment of clearly defined subacromial pain: a systematic review of randomised controlled trials. Br J Sports Med. 2016 Sep;50(18):1124-34. doi: 10.1136/bjsports-2015-095771. Epub 2016 Jun 10. PMID 27288517
- [Background] Bjornsson Hallgren HC, Adolfsson LE, Johansson K, Oberg B, Peterson A, Holmgren TM. Specific exercises for subacromial pain. Acta Orthop. 2017 Dec;88(6):600-605. doi: 10.1080/17453674.2017.1364069. Epub 2017 Aug 16. PMID 28812398
- [Background] Dahlberg LE, Dell'Isola A, Lohmander LS, Nero H. Improving osteoarthritis care by digital means - Effects of a digital self-management program after 24- or 48-weeks of treatment. PLoS One. 2020 Mar 4;15(3):e0229783. doi: 10.1371/journal.pone.0229783. eCollection 2020. PMID 32130276
- [Background] Cottrell MA, Galea OA, O'Leary SP, Hill AJ, Russell TG. Real-time telerehabilitation for the treatment of musculoskeletal conditions is effective and comparable to standard practice: a systematic review and meta-analysis. Clin Rehabil. 2017 May;31(5):625-638. doi: 10.1177/0269215516645148. Epub 2016 May 2. PMID 27141087
- [Background] Seron P, Oliveros MJ, Gutierrez-Arias R, Fuentes-Aspe R, Torres-Castro RC, Merino-Osorio C, Nahuelhual P, Inostroza J, Jalil Y, Solano R, Marzuca-Nassr GN, Aguilera-Eguia R, Lavados-Romo P, Soto-Rodriguez FJ, Sabelle C, Villarroel-Silva G, Gomolan P, Huaiquilaf S, Sanchez P. Effectiveness of Telerehabilitation in Physical Therapy: A Rapid Overview. Phys Ther. 2021 Jun 1;101(6):pzab053. doi: 10.1093/ptj/pzab053. PMID 33561280
- [Background] Gava V, Ribeiro LP, Barreto RPG, Camargo PR. Effectiveness of physical therapy given by telerehabilitation on pain and disability of individuals with shoulder pain: A systematic review. Clin Rehabil. 2022 Jun;36(6):715-725. doi: 10.1177/02692155221083496. Epub 2022 Mar 1. PMID 35230167
- [Background] Janela D, Costa F, Molinos M, Moulder RG, Lains J, Francisco GE, Bento V, Cohen SP, Correia FD. Asynchronous and Tailored Digital Rehabilitation of Chronic Shoulder Pain: A Prospective Longitudinal Cohort Study. J Pain Res. 2022 Jan 8;15:53-66. doi: 10.2147/JPR.S343308. eCollection 2022. PMID 35035234
- [Background] Cieza A, Causey K, Kamenov K, Hanson SW, Chatterji S, Vos T. Global estimates of the need for rehabilitation based on the Global Burden of Disease study 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2021 Dec 19;396(10267):2006-2017. doi: 10.1016/S0140-6736(20)32340-0. Epub 2020 Dec 1. PMID 33275908
- [Derived] Worner T, Sirard P, Nero H, Horder H, Misini Ignjatovic M, Eek F. Changes in pain and disability in patients with shoulder pain after three months of digitally delivered exercise and patient education. J Rehabil Med. 2023 Nov 14;55:jrm9415. doi: 10.2340/jrm.v55.9415. PMID 38835146